CLINICAL TRIAL: NCT04434144
Title: A Comparative Observational Study on Ivermectin and Hydroxychloroquine on the COVID19 Patients in Bangladesh
Brief Title: A Comparative Study on Ivermectin and Hydroxychloroquine on the COVID19 Patients in Bangladesh
Status: Completed | Type: Observational
Sponsor: Upazila Health & Family Planning Officer's (UHFPO) Office, Chakoria, Cox's Bazar (Other Government)
Responsible Party: Principal Investigator, Abu Taiub Mohammed Mohiuddin Chowdhury, Doctoral Resident, First Affiliated Hospital Xi'an Jiaotong University
Other Study IDs: 10000918
Record Dates: First submitted 2020-06-09; First posted 2020-06-16 (Actual); Last update posted 2020-06-16 (Actual); Status verified 2020-06

CONDITIONS: Ivermectin; Hydroxychloroquine; COVID19
Keywords: Ivermectin; Hydroxychloroquine; COVID19; Bangladesh; SARS-CoV-2
MeSH Terms: conditions — COVID-19 | interventions — Ivermectin; Doxycycline; Hydroxychloroquine; Azithromycin

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 5 Days
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (2):
- Group A:: Ivermectin 200µgm/kg single dose + Doxycycline 100mg BID for 10days
  Interventions: Drug: Ivermectin + Doxycycline
- Group B: Hydroxychloroquine 400mg first day then 200mg BID for 9days + Azithromycin 500mg daily for 5Days.
  Interventions: Drug: Hydroxychloroquine + Azithromycin

INTERVENTIONS:
Drug: Ivermectin + Doxycycline — SARS-CoV-2 infection was confirmed by RT PCR in every case. For group A, Ivermectin 200mcg/kg single dose and Doxycycline 100mg BID for 10 days were given. For group B, Hydroxychloroquine 200mg BID for 10 days and Azithromycin 500mg single daily dose for 5days was given. Before advising the contraindications and possible adverse effect and drug interactions were kept in consideration. Incase of asymptomatic patients, repeat sample collection (nasopharyngeal and throat swab) for PCR was done on 5th day. For the symptomatic patients, this duration was on the 3rd nonsymptomatic day from the first day of drug intake. In the case of positive PCR, the test was repeated after 2days and onward.
  Groups: Group A:
Drug: Hydroxychloroquine + Azithromycin — SARS-CoV-2 infection was confirmed by RT PCR in every case. For group B, Hydroxychloroquine 400mg first day then 200mg BID + Azithromycin 500mg BID for 5 days were given. For group B, Hydroxychloroquine 200mg BID for 10 days and Azithromycin 500mg single daily dose for 5days was given. Before advising the contraindications and possible adverse effect and drug interactions were kept in consideration. Incase of asymptomatic patients, repeat sample collection (nasopharyngeal and throat swab) for PCR was done on 5th day. For the symptomatic patients, this duration was on the 2nd nonsymptomatic day from the first day of drug intake. In the case of positive PCR, the test was repeated after 2days and onward.
  Groups: Group B

SUMMARY:
COVID19 is a worldwide pandemic. Hence SARS-CoV-2 is a novel virus; there is no specific medication against it. Like other countries of the world, Bangladesh is also struggling in the case of treatment of this disease. Besides antiviral drugs other existing drugs like Hydroxychloroquine, Chloroquine, and recently Ivermectin has been used for the treatment of mild to moderate cases of COVID19 disease. Till now Hydroxychloroquine has shown a good effect. Recently anti-parasitic drug Ivermectin was found highly effective in an in-vitro study against SARS-CoV-2. This study is aimed to evaluate the efficacy of Ivermectin and Hydroxychloroquine as a combination therapy with antibiotics (Doxycyclin and Azithromycin) and compare the recovery period of these two drugs applied as core monotherapy.

DETAILED DESCRIPTION:
This study was done from May 2nd to June 5th, 2020. The investigators included 181 patients who were tested positive for SARS-CoV-2 infection by RT PCR presented and the sample collected at Chokoria Upazila Health Complex, Cox's Bazar; Bangladesh. The PCR analysis of the collected sample was done at Cox's Bazar Medical College. Each of the participants was examined carefully to find out the details of the disease symptoms, history, comorbid condition, and associated complaints. Patients with severe comorbid conditions like severe Bronchial asthma, COPD exacerbation, severe ischemic heart disease, uncontrolled diabetes mellitus, advanced renal and hepatic disease, carcinoma, hospitalized and Immuno-compromised patients were not included in this study. 42 patients had comorbid conditions (some required hospitalization) that might affect the recovery time; 14 patients were unwilling to participate in the study and 9 participants did not show-up (3 from group A and 6 from group B) for follow up sample collection so these were excluded. Following exclusion 116 patients were included with mild to moderate degree of illness with normal or near-normal chest radiograph and Oxygen Saturation more than 95% were included in this study. All the patients enrolled in the study were treated as an outpatient protocol.

For the study Perouse the participants were divided into two groups as follows:

Group A (n=60): Ivermectin 200µgm/kg single dose + Doxycycline 100mg BID for 10days.

Group B (n=56): Hydroxychloroquine 400mg first day then 200mg BID for 9days + Azithromycin 500mg daily for 5Days.

Besides the above, symptomatic treatment for fever, headache, cough, myalgia, and other complaints were given accordingly. Participants were advised for self-isolation, proper nutrition, hydration, and a sanitary environment. Treatment outcomes were evaluated on every 2days starting from the 5th day (Asymptomatic patients) or the 2nd non-symptomatic day from the first day of the drug intake by PCR study of nasopharyngeal and throat swab in each group. Regular contacts were maintained to find out the adverse or side effects of the therapy. Informed consent was obtained in every case.

ELIGIBILITY:
Inclusion Criteria:

* COVID19 patients confirmed bt RT PCR at Chokoria Upazila Health Complex, Cox's Bazar; Bangladesh.
* Patients with mild to moderate degree of illness.
* Patients with normal or near-normal chest radiograph
* Patients with oxygen Saturation more than 94% who fit the outpatient treatment protocol.

Exclusion Criteria:

* Patients with severe uncontrolled comorbid conditions. (Bronchial asthma, COPD exacerbation, ischemic heart disease, uncontrolled diabetes mellitus, advanced renal and hepatic disease, carcinoma, hospitalized, Immuno-compromised patients)
* BMI>30
* Contraindication / possible drug interaction with Ivermectin and Hydroxychloroquine.

Ages: 16 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: The total number of patients was 116; male 84 and female 26, age 16 to 80years, mean age 33.94years.
  Group A (Ivermectin + Doxycyclin): male 43 (71.67%), female 17 (28.33%), age 35.72 ± 15.1 years. Male 37and, female 32.88 years.
  Group B (Hydroxychloroquine + Azithromycin): male 47 (83.93%), female 9(16.07%), age 31.91years. Male 31.35, and female 34.5 years.
Sampling Method: Probability Sample
Enrollment: 116 (Actual)
Dates: Start 2020-05-02 (Actual); Primary Completion 2020-06-05 (Actual); Study Completion 2020-06-05 (Actual)

PRIMARY OUTCOMES:
Number of participants with "treatment success" determine by a negative RT PCR for COVID19. | 02/05/2020 to 05/06/2020
  Treatment outcomes of the COVID19 positive participants will be evaluated on the 5th day in case of an asymptomatic participant; in case of the symptomatic participant, on the 2nd non-symptomatic day onward from the first day of the drug intake by PCR study of nasopharyngeal and throat swab. In the case of still positive PCR, the swab will be collected from the participants after every 2days until the status is negative. A negative PCR is a count of treatment success in each case. The duration (in days) from the first day of drug intake to the negative PCR is the recovery period. Participants who require hospitalization or decease due to the disease progression during the treatment will count as treatment failure.
Number of participants with "adverse effects" determined by the existence of the pharmacological side effects of the particular drug during treatment. | 02/05/2020 to 05/06/2020
  The adverse effect will define as the symptoms expressed by the participants following the starting of the treatment other than the disease symptoms, those are within the proven/enlisted pharmacological side effects of the particular drug therapy. Adverse effects will be evaluated by communication on phone or during the follow up sample collection by detailed history taking. The degree of symptoms will be noted as continuous/occasional and mild/ moderate/severe.

CONTACTS AND LOCATIONS:
Overall Officials: Abu Taiub Mohammed Mohiuddin Chowdhury, MBBS, MD, Study Director — First Affiliated Hospital Xi'an Jiaotong University; Mohammad Shahbaz, MBBS, MCPS, Study Chair — Upazila Health & Family Planning Officer's (UHFPO) Office, Chakoria, Cox's Bazar
Locations (1):
- Chakoria Upazilla Health Complex, Cox’s Bāzār, Bangladesh

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Patri A, Fabbrocini G. Hydroxychloroquine and ivermectin: A synergistic combination for COVID-19 chemoprophylaxis and treatment? J Am Acad Dermatol. 2020 Jun;82(6):e221. doi: 10.1016/j.jaad.2020.04.017. Epub 2020 Apr 10. No abstract available. PMID 32283237
- [Background] Zhou D, Dai SM, Tong Q. COVID-19: a recommendation to examine the effect of hydroxychloroquine in preventing infection and progression. J Antimicrob Chemother. 2020 Jul 1;75(7):1667-1670. doi: 10.1093/jac/dkaa114. PMID 32196083
- [Background] Yao X, Ye F, Zhang M, Cui C, Huang B, Niu P, Liu X, Zhao L, Dong E, Song C, Zhan S, Lu R, Li H, Tan W, Liu D. In Vitro Antiviral Activity and Projection of Optimized Dosing Design of Hydroxychloroquine for the Treatment of Severe Acute Respiratory Syndrome Coronavirus 2 (SARS-CoV-2). Clin Infect Dis. 2020 Jul 28;71(15):732-739. doi: 10.1093/cid/ciaa237. PMID 32150618
- [Background] Lv C, Liu W, Wang B, Dang R, Qiu L, Ren J, Yan C, Yang Z, Wang X. Ivermectin inhibits DNA polymerase UL42 of pseudorabies virus entrance into the nucleus and proliferation of the virus in vitro and vivo. Antiviral Res. 2018 Nov;159:55-62. doi: 10.1016/j.antiviral.2018.09.010. Epub 2018 Sep 26. PMID 30266338
- [Background] Caly L, Druce JD, Catton MG, Jans DA, Wagstaff KM. The FDA-approved drug ivermectin inhibits the replication of SARS-CoV-2 in vitro. Antiviral Res. 2020 Jun;178:104787. doi: 10.1016/j.antiviral.2020.104787. Epub 2020 Apr 3. PMID 32251768